CLINICAL TRIAL: NCT06344390
Title: Effect of Pentoxifylline on Cognitive Impairment After Ischemic Stroke and Its Mechanism of Brain Electricity and Brain Metabolism
Brief Title: Effect of Pentoxifylline on Cognitive Impairment After Ischemic Stroke
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Bing Han, associate chief physician, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210327
Record Dates: First submitted 2023-12-25; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pentoxifylline (Experimental): Pentoxifylline
  Interventions: Drug: Pentoxifylline
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Pentoxifylline — Take pentoxifylline 0.4 g twice daily
  Other Names: CSPC Pharmaceutical Group
  Arms: Pentoxifylline

SUMMARY:
Pentoxifylline can improve cognitive impairment after ischemic stroke, possibly by improving the level of cerebral blood flow, affecting the content of blood oxygen and metabolic substances in the brain, and then playing a protective role in the transmission of nerve electrical signals, and ultimately improving cognitive function. The patients with cognitive impairment and non-dementia PSCIND after ischemic stroke were randomly divided into two groups. In addition to the basic drugs of ischemic stroke, the patients were given pentothemine sustained release tablets and blank control respectively to observe the effects of pentothemine on cognitive function and neuronal electrical signals in the patients with ischemic PSCIND. It is expected to explore the possible internal biological mechanism by using transcranial Doppler, oxygen-dependent functional magnetic resonance imaging and craniocerebral magnetic resonance pop analysis. Finally, statistical correlation analysis was used to elucidate the specific mechanism of pentoxifylline in improving cognitive function of non-dementia patients with cognitive impairment after ischemic stroke.

DETAILED DESCRIPTION:
Pentoxifylline can improve cognitive impairment after ischemic stroke, possibly by improving the level of cerebral blood flow, affecting the content of blood oxygen and metabolic substances in the brain, and then playing a protective role in the transmission of nerve electrical signals, and ultimately improving cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Han Chinese, age 40-80 years old, male and female, right-handed;
* The diagnosis is consistent with the Expert Consensus on the Management of Cognitive Impairment after Stroke 2021;
* NIHSS score 1-15 points;
* Daily Living Ability Scale (ADL) ≥75 score;
* The Informed consent signed by the patient or his legal representative

Exclusion Criteria:

* Can not cooperate with the examination (including neuropsychological tests and scale assessment);
* There were memory disorders, dementia with lewy bodies and frontotemporal dementia before the onset of stroke events;
* There were definite infectious diseases 2 weeks before admission; Have a serious mental illness, previous history of cancer, alcohol or drug abuse;
* Use of drugs that may affect cognitive function, including sedatives, anti-anxiety drugs, hypnotics, nootropic drugs, and cholinoid drugs;
* Can not accept brain MRI examination

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pentoxifylline can improve cognitive impairment after ischemic stroke | 3 months
  The Montreal Cognitive Assessment, MoCA: A Brief Screening Tool For Mild Cognitive Impairment.If the score is less than 26 points, it is considered to have cognitive impairment.Patient scores get higher after 3 months, we think pentoxifylline can improve cognitive impairment after ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Jiaying Rong, master, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- BHan, Shijiazhuang, China

IPD SHARING:
Plan to Share IPD: No